CLINICAL TRIAL: NCT06275217
Title: The Effects of a Mindful Yoga Program on Mood Symptoms and Stress for Postpartum Women With Depressive Symptoms: a Randomized Controlled Clinical Trial
Brief Title: Mindful Yoga for Postpartum Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LIN Jingxia Jessie, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HMRF17182481
Record Dates: First submitted 2024-01-17; First posted 2024-02-23 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Mood Disorders
Keywords: Yoga; Mindfulness-based; Postpartum depression; mood symptoms
MeSH Terms: conditions — Mood Disorders; Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful yoga group (Experimental): The participants in experimental group will receive a 10-week mindfulness-based yoga program, one session per week with 1.5 hours in each session.
  Interventions: Behavioral: Mindfulness-based yoga program
- Psychoeducation group (Active Comparator): The participants in the psychoeducation group will receive a 10-week psychoeducation program, one session per week with 1.5 hours in each session.
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Behavioral: Mindfulness-based yoga program — The intervention includes mindfulness-based components and yoga practice. Once a week for 10 weeks, with 1.5 hours in each session (30 minutes mindfulness-based practice and 1 hour yoga practice). A well-trained research personnel will facilitate the mindfulness-based section, and a qualified yoga instructor will facilitate the yoga section.
  Arms: Mindful yoga group
Other: Psychoeducation — Knowledge of perinatal mental health, stress-related management, postnatal nutrition, exercise habit and sleep hygiene will be provided to the participants in the psychoeducation group. It is a group-based intervention delivered in hybrid mode including face-to-face and online group-based class. Once a week for 10 weeks, with 1.5 hour in each session.
  Arms: Psychoeducation group

SUMMARY:
This is a parallel-group randomized controlled trial. A total of 198 postpartum women with depressive symptoms (EPDS scores≥8 at baseline) will be recruited and randomized into two groups: 10-week mindful yoga intervention and 10-week psychoeducation program. Clinical assessment of depression, self-report questionnaires and salivary cortisol tests will be performed at baseline, after 10-week intervention, and at 6-month and 12-month follow-ups. The investigators expected that the mindful yoga intervention will reduce depression after 10 weeks compared to psychoeducation. The mindful yoga intervention will further reduce anxiety, stress, improve quality of life and sleep, and steepen diurnal cortisol slopes. These effects will be maintained for at least six months.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women aged 18-60 years old.
* The scores of EPDS ≥ 10.
* At least 6 week and up to 1 year after childbirth.
* Giving birth to a single full-term healthy baby (gestation between 37-41 weeks, body weight > 2.5kg, APGAR score at 5 minutes > 7).
* Fewer than 10 hours of yoga/Qi gong/Tai Chi or mindfulness/meditation practice in the previous 3 months.

Exclusion Criteria:

* Severe complications after delivery, or their infants are admitted to NICU.
* Regular psychiatric follow-up.
* Currently taking antipsychotic drugs.
* Known pragnancy, or other contraindications to physical exercise (e.g., wound healing situation) according to the body examination by O&G clinicians at 6 weeks after delivery.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Postpartum women with depression.
Enrollment: 198 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale | Baseline, 10 weeks, 6 months and 1 year follow-ups.
  Measures postnatal depression. Each item scores 0-3, and the total score ranges from 0 to 30. Higher score means worse depressive symptoms.

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale-Depression | Baseline, 10 weeks, 6 months and 1 year follow-ups.
  Measures depressive symptoms. Each item scores 0-3, the total score for depression ranges from 0 to 21. Higher score means worse symptoms of depression.
Depression Anxiety Stress Scale-Anxiety | Baseline, 10 weeks, 6 months and 1 year follow-ups.
  Measures anxiety symptoms. Each item scores 0-3, the total score for anxiety ranges from 0 to 21. Higher score means worse symptoms of anxiety.
Depression Anxiety Stress Scale-Stress | Baseline, 10 weeks, 6 months and 1 year follow-ups.
  Measures stress symptoms. Each item scores 0-3, the total score for stress ranges from 0 to 21. Higher score means worse symptoms of stress.
Pittsburgh Sleep Quality Index | Baseline, 10 weeks, 6 months and 1 year follow-ups.
  Measures sleep quality. There are 8 components scores, and each component score ranges from 0 to 3. Higher score means worse sleep quality.
36 Item-Short Form Health Survey Questionnaire | Baseline, 10 weeks, 6 months and 1 year follow-ups.
  Measures quality of life including physical and mental health. Each item scores 0-100. There are eight subscores ranging from 0 to 100. Higher score means better quality of life.
Five Facet Mindfulness Questionnaire | Baseline, 10 weeks, 6 months and 1 year follow-ups.
  Measures the level of mindfulness ability. Each item scores 1-5, and the total score ranges from 42 to 210. Higher score means better mindfulness ability.
Pregnancy Symptom Inventory | Baseline, 10 weeks, 6 months and 1 year follow-ups.
  Measures physical pain and fatigue of postpartum women. Each item scores 0-3. The total score ranges from 0 to 24. Higher score means worse pregnancy symptoms.
Cortisol concentration level | Baseline and 10 weeks (post-intervention).
  Measures salivary cortisol concentration at baseline and post-intervention. Higher concentration means higher level of stress and depression.
Physical fitness | Baseline and 10 weeks (post-intervention).
  6-minute walking test is used for physical fitness measure. The total distance walked during 6 minutes is recorded. Higher score means better fitness.
Balance | Baseline and 10 weeks (post-intervention).
  Single-leg standing test is used to measure the balance. The time to keep the posture is recorded. Higher score means better balance ability.

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Lin, PhD, Study Chair — Department of Rehabilitation Sciences, The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong